CLINICAL TRIAL: NCT03041883
Title: Corneal Collagen Crosslinking to Increase the Resistance of the Graft Used as a Support for the Boston Keratoprosthesis Type I Against Corneal Melting
Brief Title: Corneal Collagen Crosslinking to Increase the Resistance of the Support Graft of the KPro Type I Against Corneal Melting
Acronym: CXL-KPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE14.362
Record Dates: First submitted 2017-01-25; First posted 2017-02-03 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Corneal Melting in Boston Keratoprosthesis Type I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kpro with crosslinked graft-support (Experimental): Patient will receive a crosslinked corneal graft-support for the KPro type I. Under sterile conditions, the corneo-scleral button will be inspected, then placed on an artificial anterior chamber. The epithelium of the donor will be removed mechanically. Then one drop of riboflavin 0.1%/dextran 20% will be applied to 3 minutes on the de-epithelialized cornea for 15 minutes. Then, the source of ultraviolet A (UVA) will be irradiating the cornea for 30 minutes with a wavelength of 370 nanometer(nm) length with 5.4 joules(J)/ square centimeter (cm2) and 3 milliwatts(mW)/cm2. Meanwhile, the instillation of a drop of 0.1% riboflavin/dextran 20% continues every 5 minutes. Goggles against UVA are mandatory. The crosslinked graft-support will be forwarded to the surgeon according to standard procedure.
  Interventions: Procedure: Crosslinking with riboflavin of the corneal graft-support
- KPro with normal graft-support (Active Comparator): Patient wil receive a normal graft-support for the KPro type I. Under sterile conditions, the corneo-scleral button will be inspected, then placed on an artificial anterior chamber. The epithelium of the donor will be removed mechanically. Then, one drop of riboflavin 0.1% / dextran 20% will be applied to 30 secondes for 5 minutes on the de-epithelialized cornea.The minimally manipulated normal graft-support will be forwarded to the surgeon according to standard procedure.
  Interventions: Procedure: De-epithelisation of the corneal graft support with instillation of riboflavin

INTERVENTIONS:
Procedure: Crosslinking with riboflavin of the corneal graft-support — Corneal graft support for the KPro will be crosslinked and used with the standard surgical technique
  Arms: Kpro with crosslinked graft-support
Procedure: De-epithelisation of the corneal graft support with instillation of riboflavin — Corneal graft-support will be de-epithelialized and soaked with riboflavin and then used with the standard surgical technique
  Arms: KPro with normal graft-support

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of the corneal collagen crosslinking with riboflavin and ultraviolet A in aim to increase the resistance of the graft used as a support for the Boston keratoprosthesis (KPro) type I against corneal melting (keratolysis or sterile necrosis).

DETAILED DESCRIPTION:
The Boston type 1 keratoprosthesis (KPro) is an artificial cornea that restores the clarity of the visual axis. It is indicated in patients for whom conventional corneal transplantation offers a very low probability of success. Several innovations have led to improved outcomes following implantation of a KPro. However, retention of the KPro varies between 83 and 100% in the most recent series. The extrusion of the KPro is usually caused by the melting of the corneal tissue (keratolysis or sterile necrosis) used as a support.

This corneal melting is mediated by enzymes from the class of the matrix metalloproteinases (MMP). Several different types of insults may lead to an excess of these enzymes. Chronic inflammation of the ocular surface is undoubtedly the best recognized risk factor. Indeed, autoimmune diseases such as Stevens-Johnson syndrome, Lyell syndrome (toxic epidermal necrolysis, TENS) and mucous membrane pemphigoid, has the highest rate of corneal melting post KPro. Moreover, the development of a retroprosthetic membrane has recently been recognized as a risk factor for melting. Furthermore, the dryness of the corneal epithelium, due to insufficient tear production or an alteration of the blink reflex of the eye, can also lead to an overexpression of MMP. Finally, infectious keratitis can lead to significant thinning of the corneal tissue, even once the infectious process is resolved.

Corneal collagen cross-linking is a technique approved by Health Canada for strengthening the biomechanical properties of the cornea. The crosslinked corneas become more resistant to collagenase and other MMP. The use of a crosslinked corneal graft as a support for the KPro is an interesting approach to the prevention of corneal melting.

A prospective, randomized, controlled and double-blind study will be conducted with patients receiving a Kpro at the Centre Hospitalier de l'Université de Montréal. Forty patients will be randomized into two groups, half will receive KPro in a crosslinked graft-support, while the other half will receive a usual graft-support. Patients will be met by their surgeon to discuss the risks, benefits of the KPro type I and alternatives treatments. Patients accepting KPro surgery, will be informed of the nature and course of the study and will be offered to participate in the study. The Eye bank of Canada will manage the randomization and maintain the codes identifying the crosslinked corneas from the untreated corneas, keeping both the surgeon and the patient blinded. Randomization will be done through a free application (http://www.randomizer.org/form.htm). A series of 10 numbers will be generated. Even numbers indicate crosslinked corneas and odd numbers indicate non-crosslinked corneas. The order of the digits will increase as for each subject is enrolled in the study. The procedure for corneal collagen crosslinking will be performed at the Eye Bank of Canada in a similar procedure to the treatment for keratoconus. Under sterile conditions, the corneo-scleral button will be inspected to meet the standard of care. If the patient is randomized to the crosslinked group, then the cornea will be treated with crosslinking as described further. If the patient is randomized the control group, the cornea will not be treated with crosslink but will be deepithelialized and soaked with riboflavin drops as described further.

The surgeon will receive the graft and operate according to the standard procedure. The KPro surgery and postoperative care will be performed in the standard way and thus will be the same for both study groups. Postoperative follow will be held at 1 day, 1 week, 2 weeks, 1 month and 3 months and will continue subsequently every 2-4 months depending on the judgment of the surgeon. These visits will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination. In particular, the presence of corneal melting, leakage of aqueous humor, corneal infection and extrusion will be noted. Meanwhile, an imaging allowing quantification of the thickness of the cornea graft-support (optical coherence tomography anterior segment) will be performed at least once during the first three months postoperative. This imaging will be repeated at 1, 2 and 5 years.

The prevalence of various complications (melting, leak, infection, extrusion) will be compared between the two groups with the Fischer exact test. Also, the time between surgery and the occurrence of complications will be compared using the Student t test. Finally, survival analysis of Kaplan-Meier will be performed for 1) the occurrence of corneal melting and 2) maintaining a visual acuity greater than 20/200.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for KPro type I
* Capacity to give written consent
* Ability to be followed for the duration of the study

Exclusion Criteria:

* Participation in another interventional study
* Failure to wear a therapeutic contact lens due to abnormalities of the eyelids.
* Inability to give written consent

Contraindications to the KPro type I:

* Severe dryness with keratinization of the ocular surface
* Intraocular tumor
* Terminal glaucoma
* Inoperable retinal detachment
* Phthisis bulbi

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 1 day
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 1 week
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 2 weeks
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 1 month
  This visits will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 1 month
  An imaging allowing quantification of the thickness of the cornea graft-support (optical coherence tomography anterior segment) will be performed.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 3 months
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | Every 2-4 months depending on the judgment of the surgeon for at least 5 years
  These visits will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 1 year
  An imaging allowing quantification of the thickness of the cornea graft-support (optical coherence tomography anterior segment) will be performed.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 2 years
  An imaging allowing quantification of the thickness of the cornea graft-support (optical coherence tomography anterior segment) will be performed.
Examine whether the use of crosslinked cornea decreases the rate of corneal melting post-Kpro when compared to using a standard corneal button | 5 years
  An imaging allowing quantification of the thickness of the cornea graft-support (optical coherence tomography anterior segment) will be performed.

SECONDARY OUTCOMES:
Comparison of the rates of infectious keratitis between the groups | 1 day
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of infectious keratitis between the groups | 1 week
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of infectious keratitis between the groups | 2 weeks
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of infectious keratitis between the groups | 1 month
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of infectious keratitis between the groups | 3 months
  This visits will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of infectious keratitis between the groups | Every to 2-4 months depending on the judgment of the surgeon for at least 5 years
  These visits will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of extrusion of the KPro between the groups | 1 day
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of extrusion of the KPro between the groups | 1 week
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of extrusion of the KPro between the groups | 2 weeks
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of extrusion of the KPro between the groups | 1 month
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of extrusion of the KPro between the groups | 3 months
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the rates of extrusion of the KPro between the groups | Every to 2-4 months depending on the judgment of the surgeon for at least 5 years
  These visits will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the visual acuity between the groups | 1 day
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the visual acuity between the groups | 1 week
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the visual acuity between the groups | 2 weeks
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the visual acuity between the groups | 1 month
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the visual acuity between the groups | 3 months
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.
Comparison of the visual acuity between the groups | Every to 2-4 months depending on the judgment of the surgeon for at least 5 years
  This visit will include measurement of visual acuity and intraocular pressure and a full slit-lamp examination.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Robert, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558